CLINICAL TRIAL: NCT03619928
Title: Comparison of Dry Needle and Massotherapy on Tolerance to the Effort and Soreness of Individuals With Late Muscular Pain Induced by Exercise
Brief Title: Comparison of Dry Needle and Massotherapy on Tolerance Effort and Soreness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, ROMERO SOUZA LEÃO DE ALBERGARIA CRASTO, Principal researcher, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DN, massotherapy and DOMS
Record Dates: First submitted 2018-07-27; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: Dry needling; Massotherapy; Delayed onset muscle soreness
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Procedure in which a thin needle is used to penetrate the skin, subcutaneous tissues and muscle with the intention of mechanically stimulating the tissue without the use of an anesthetic. The physiological mechanism supporting the effects of dry needling remains to be clarified. It has been suggested that the needle works according to the pain gate control theory, indicating that one type of sensory input could be inhibited in the Central nervous system by another input
  Interventions: Device: Dry needling
- Massotherapy (Active Comparator): Among the therapeutic approaches for DOMS is massage therapy. Several authors have examined the effects of DOMS massage and indirect markers of muscle damage, such as impaired muscle function, edema and muscle changes in blood proteins.
  Interventions: Device: Massotherapy

INTERVENTIONS:
Device: Dry needling — 20 minutes through a sterile, disposable Dong Bang® needle size of 0.25X30 mm. At the moment of insertion of the needle, the therapist will perform a muscular shortening around the application site, in a pincer movement performed by the index and thumb fingers, in order to isolate the muscle fibers of the biceps brachii. Five needles will be applied to the short head brachii biceps in five points: origin, insertion, center of the muscular womb (60% of the distance from the medial acromion to the cubital fossa in the elbow line) and two points equidistant from the center 2 cm.
  Arms: Dry needling
Device: Massotherapy — A 20-minute massage will be applied to the non-dominant upper limb exercised by a therapist for the massage condition. The massage will consist of: 1) surface slip; 2) deep slip; 3) kneading; 4) friction with the thumbs; 5) friction with four fingers; 6) percussions with open and alternating hands; 7) percussions with open and simultaneous hands; 8) tapping; and 9) surface slip.
  Arms: Massotherapy

SUMMARY:
Introduction: Delayed onset muscle soreness (DOMS) is a common myogenic condition considered to be a muscle tension injury frequently observed in recreational or experienced athletes, induced in the majority of cases by eccentric and inactive exercises, the most common of which are: tension, pain and impairment muscular and have a course of typical duration of 24 hours and peak between 48 and 72 hours. Among the treatments proposed with the aim of reducing the symptoms of DOMS is massage therapy. However, dry needling is a relatively new technique that has been used in myotendinous lesions and its effects on late muscle pain have not yet been studied. Objective: To compare the impact of dry needling and massage therapy on exercise tolerance, and analgesia of sedentary individuals with late muscle pain induced by eccentric exercise. The present study is characterized as a randomized and blinded comparative study in which male sedentary individuals will be invited in which the late muscle pain will be induced through eccentric contractions and will receive different treatments: dry needling or massage therapy. The upper limb functionality, pain perception, superficial hyperemia and brachial biceps thickness will be compared through the exams: visual analogue pain scale (VAS), digital algometry, thermography, ultrasonography and isometric test.

ELIGIBILITY:
Inclusion Criteria:

not practicing physical activity BMI greater than 18 and less than 30 members of the UFPE community

Exclusion Criteria:

making use of analgesic or anti-inflammatory medications acupuncture or dry needling or massage therapy in the last 6 months report of muscle pain orthopedic neurological problems hypertension and diabetes cardiovascular or respiratory diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-08-27 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | 48 hours
  Algometry
Delayed onset muscle soreness | 48 hours
  Visual analogue scale which measures the pain and whose minimum value is zero and the maximum value is 100 millimeters. The higher value is the worse the pain.

SECONDARY OUTCOMES:
Muscle thickness | 48 hours
  Ultrassonography
Temperature | 48 hours
  Thermography
Time limit | 48 hours
  Isometric performance test

CONTACTS AND LOCATIONS:
Overall Officials: Romero SL Crasto, Esp., Principal Investigator — Master student, program in physical therapy
Locations (1):
- Romero Souza Leão de Albergaria Crasto, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No